CLINICAL TRIAL: NCT03267316
Title: An Open Label, Dose Escalation Followed by Dose Expansion, Safety and Tolerability Trial of CAN04, a Fully Humanized Monoclonal Antibody Against IL1RAP, in Subjects With Solid Malignant Tumors
Brief Title: A First-in-Human Study of CAN04 in Patients With Solid Malignant Tumors
Acronym: CANFOUR
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cantargia AB (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CAN04CLIN001; 2017-001111-36 (EudraCT Number)
Record Dates: First submitted 2017-08-24; First posted 2017-08-30 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Non Small Cell Lung Cancer; Pancreatic Ductal Adenocarcinoma; Triple Negative Breast Cancer; Colorectal Cancer
Keywords: First-in-Human; Phase 1; Phase 2; Antibody, Monoclonal; IL1RAP; Safety; Tolerability; Cancer; Solid tumor; Malignant; Dose escalation; Dose expansion; CAN04; Immunoglobulin; Clinical Trial; Infusion; Antineoplastic; Anticancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Triple Negative Breast Neoplasms; Colorectal Neoplasms; Neoplasms | interventions — Cisplatin; Gemcitabine; 130-nm albumin-bound paclitaxel; Carboplatin; Pemetrexed

STUDY DESIGN:
Intervention Model Description: Part I of the study is designed to define the Maximum Tolerated Dose/ Recommended Phase 2 Dose (MTD/RP2D) of CAN04 in subjects with relapsed or refractory Non-Small Cell Lung Cancer (NSCLC), Pancreatic Ductal Adenocarcinoma (PDAC), Triple Negative Breast Cancer (TNBC) or Colorectal Cancer (CRC). [Completed December 2018]
  Part II consists of seven treatment arms and aims to establish the safety and tolerability of CAN04 as monotherapy and in combination with the standard of care in subjects with NSCLC or PDAC, as well as to investigate early signs of efficacy [Enrollment to all arms completed].
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Dose escalation (Experimental): Cohorts of 3 subjects will receive once weekly (Q1W) treatment with CAN04. The Dose Limiting Toxicity (DLT) observation period for each dose level will be the first 21 days of treatment with CAN04. [Completed December 2018]
  Interventions: Biological: CAN04
- Monotherapy (Q1W) (Experimental): Subjects with either PDAC or NSCLC, will receive treatment with CAN04 monotherapy once weekly (Q1W).
  Interventions: Biological: CAN04
- Monotherapy (Q1W/Q2W) (Experimental): Subjects with either PDAC or NSCLC, will receive treatment with CAN04 monotherapy once weekly (Q1W) for the first 6 weeks followed by treatment every second week (Q2W).
  Interventions: Biological: CAN04
- Combination - NSCLC (NCG) (Experimental): Subjects with NSCLC will receive treatment with CAN04 once weekly (Q1W) for the first 6 weeks followed by treatment every second week (Q2W) in combination with standard-of-care therapy (cisplatin/gemcitabine).
  Interventions: Biological: CAN04; Drug: Cisplatin; Drug: Gemcitabine
- Combination - PDAC (Experimental): Subjects with PDAC will receive treatment with CAN04 once weekly (Q1W) for the first 6 weeks followed by treatment every second week (Q2W) in combination with standard-of-care therapy (nab-paclitaxel/gemcitabine).
  Interventions: Biological: CAN04; Drug: Gemcitabine; Drug: Nab-paclitaxel
- Combination - PDAC (1 mg/kg) (Experimental): Subjects with PDAC will receive CAN04 on Day 1 and 15 in cycles of 28 days in combination with standard-of-care therapy (nab-paclitaxel/gemcitabine). During first cycle CAN04 also to be administered on Day 8.
  Interventions: Biological: CAN04; Drug: Gemcitabine; Drug: Nab-paclitaxel
- Combination - PDAC (2,5 mg/kg) (Experimental): Subjects with PDAC will receive CAN04 on Day 1 and 15 in cycles of 28 days in combination with standard-of-care therapy (nab-paclitaxel/gemcitabine). During first cycle CAN04 also to be administered on Day 8.
  Interventions: Biological: CAN04; Drug: Gemcitabine; Drug: Nab-paclitaxel
- Combination - non-squamous NSCLC (NCP) (Experimental): Subjects with non-squamous NSCLC will receive CAN04 on Day 1 and 8 in cycles of 21 days in combination with standard-of-care therapy (carboplatin/pemetrexed).
  Interventions: Biological: CAN04; Drug: Carboplatin; Drug: Pemetrexed

INTERVENTIONS:
Biological: CAN04 — A fully humanized monoclonal immunoglobulin G1 (IgG1) antibody (hmAb) in aqueous solution administered by i.v. infusion.
Drug: Cisplatin — Standard of care treatment
  Arms: Combination - NSCLC (NCG)
Drug: Gemcitabine — Standard of care treatment
  Arms: Combination - NSCLC (NCG); Combination - PDAC; Combination - PDAC (1 mg/kg); Combination - PDAC (2,5 mg/kg)
Drug: Nab-paclitaxel — Standard of care treatment
  Arms: Combination - PDAC; Combination - PDAC (1 mg/kg); Combination - PDAC (2,5 mg/kg)
Drug: Carboplatin — Standard of care treatment
  Arms: Combination - non-squamous NSCLC (NCP)
Drug: Pemetrexed — Standard of care treatment
  Arms: Combination - non-squamous NSCLC (NCP)

SUMMARY:
This study will evaluate the safety, tolerability, and preliminary antitumor activity of CAN04 both as a monotherapy and in combination with standard of care treatment in subjects with solid cancer tumors.

Following completion of the first part, the dose escalation cohorts, and determination of maximum tolerated dose or recommended phase 2 dose (MTD/RP2D), safety and tolerability will be further evaluated in an expanded cohort of subjects with pancreatic or lung cancer, as monotherapy or in combination with the standard of care treatment and to identify the RP2D of CAN04 in combination with standard of care. In addition, early signs of efficacy during treatment with CAN04 will be investigated.

DETAILED DESCRIPTION:
CAN04 is a first-in-class fully humanized and ADCC enhanced monoclonal antibody, targeting the Interleukin 1 Receptor Accessory Protein (IL1RAP).

The CAN04 strategy is to attack the IL1RAP target molecule using an effective antibody-based cancer treatment. In preclinical (in vitro and in vivo) studies, CAN04 has shown two distinct mechanisms of action:

1. By blocking the intracellular signals from the IL1RAP target molecule, thereby impairing the cancer cells' ability to secrete tumor stimulating cytokines, in turn reducing tumor inflammation and tumor progression.
2. Through antibody dependent cellular cytotoxicity (ADCC) against IL1RAP expressing tumor cells where CAN04 stimulates natural killer (NK) cells to attack the tumor cells.

The study is a combined phase 1/2a, open-label, dose-escalation followed by dose expansion, safety and tolerability clinical trial, in patients with relapsed or refractory solid tumors. It consists of two parts.

In Part I (Dose Escalation - DE), the intention is to include patients with any of the four solid tumor types: Non-Small Cell Lung Cancer (NSCLC), Pancreatic Ductal Adenocarcinoma (PDAC), Triple Negative Breast Cancer (TNBC) or Colorectal Cancer (CRC). In this part of the study safety and tolerability will be documented and the MTD/ RP2D will be determined. Patients will stay on CAN04 treatment until disease progression, unacceptable toxicity, or discontinuation for any other reason. [Completed December 2018]

In Part II (Expansion Cohort - EC), safety and tolerability will be further evaluated in an expanded cohort of subjects with PDAC or NSCLC to identify RP2D of CAN04 in combination with standard of care. In addition, early signs of efficacy during treatment with CAN04 will be investigated, as monotherapy or in combination with the standard of care.

Patients will stay on treatment until disease progression, unacceptable toxicity, or discontinuation for any other reason. [Enrollment to all arms completed]

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 year.
2. Measurable disease in accordance to iRECIST by computed tomography (CT) or magnetic resonance imaging (MRI) scan, no more than 6 weeks prior to screening.
3. At least 4 weeks since the last dose of radiation therapy, immunotherapy, or surgery; at least 6 weeks for therapy which is known to have delayed toxicity; at least 4 weeks since treatment with biologic/targeted therapies.
4. Eastern Cooperative Oncology Group (ECOG) performance status ≤1.
5. Histologically or cytologically confirmed diagnosis of unresectable stage III or stage IV squamous or non-squamous NSCLC (applicable Part II, Combination - NSCLC (NCG) arm only).

   * Subjects must be eligible to receive first line standard chemotherapy regimen with cisplatin/gemcitabine or a second line standard chemotherapy regimen with cisplatin/gemcitabine after relapsing from first line with pembrolizumab monotherapy.
   * Subjects with actionable mutations (EGFR, ALK, ROS) can be enrolled if they have previously progressed to all approved standard of care targeted therapies and the next line of standard therapy is a platinum doublet.
6. Histologically or cytologically confirmed diagnosis of unresectable stage III or stage IV non-squamous NSCLC (applicable Part II, Combination - non-squamous NSCLC NCP arm only).

   * Subjects must be eligible to receive first line standard chemotherapy regimen with carboplatin/pemetrexed or a second line standard chemotherapy regimen with carboplatin/pemetrexed after relapsing from first line with pembrolizumab monotherapy.
   * Subjects with actionable mutations (EGFR, ALK, ROS) can be enrolled if they have previously progressed to all approved standard of care targeted therapies and the next line of standard therapy is a platinum doublet.
7. Newly diagnosed, treatment naїve, histologically confirmed, unresectable, locally advanced or metastatic (stage III or stage IV) PDAC (applicable Part II, Combination - PDAC arms only).

   * Subjects must be eligible to receive treatment with nab-paclitaxel and gemcitabine.

Exclusion Criteria:

1. Subjects receiving live vaccination, etanercept or other TNF-α inhibitors or any other investigational agents during or just prior to (within 28 days of first study drug administration) participation in this study.
2. Clinical evidence of an active metastatic second malignancy.
3. Subjects with a life expectancy <12 weeks.
4. Uncontrolled or significant cardiovascular disease defined as New York Heart Association Classification III, or IV.
5. Immunocompromised subject currently receiving systemic therapy.
6. Other medical conditions that in the opinion of the investigator disqualify the subject for inclusion.
7. Applicable Part II, Combination - NSCLC (NCG and NCP) arms only

   * Prior lines of treatment with anti-cancer medication other than pembrolizumab administered as 1st line.
   * Known tumor EGFR mutation, unless contraindication to EGFR-directed therapy or if the subject has progressed to all approved anti-EGFR therapies.
   * Known tumor ALK rearrangements, unless contraindication to ALK-directed therapy or ALK-directed therapy not available or if the subject has progressed to all approved anti-EGFR therapies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-03-14 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | From the first dose until the last subject has completed their end of trial visit or the last enrolled subject has completed 6 months of treatment, whichever occurs first
  The incidence of Grade 3 or higher adverse events (AEs) related to CAN04 administration and according to the National Cancer Institute - Common Terminology Criteria for Adverse Events (CTCAE, version 4.03).

SECONDARY OUTCOMES:
Maximum concentration (Cmax) | 5 weeks
  Maximum plasma concentration of CAN04
Terminal half-life (t1/2) | 5 weeks
  Terminal half-life of CAN04
Clearance (CL) | 5 weeks
  Plasma clearance of CAN04
Apparent volume of distribution during the terminal phase (VZ) | 5 weeks
  Apparent volume of distribution of CAN04 during the terminal phase
Area under the curve from time 0 to infinity (AUC0-∞) | 5 weeks
  Area under the plasma concentration curve from time 0 to infinity
Anti-drug antibodies (ADA) against CAN04 | Through study completion, an average of 6 months
  Immunogenicity of CAN04 after repeated administrations, assessed by ADA titers in serum.
Preliminary signs of efficacy as assessed by tumor response | One year
  Tumor response (irRC Part I Part II Monotherapy arms; iRECIST Part II Combination arms)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Awada, Professor, Principal Investigator — Jules Bordet Institute, Brussels, Belgium
Locations (25):
- Austria (2):
  - Landeskrankenhaus Salzburg, Salzburg
  - Medizinische Universität Wien, Vienna
- Belgium (3):
  - Institut Jules Bordet, Brussels
  - University Hospital Gasthuisberg, Leuven
  - CHU de Liège, Liège
- Denmark (4):
  - Aalborg University Hospital, Aalborg
  - Rigshospitalet, Department of Oncology, Copenhagen
  - Herlev og Gentofte Hospital, Herlev
  - Odense University Hospital, Odense
- Estonia (2):
  - East Tallinn Central Hospital, Tallinn
  - Tartu University Hospital, Tartu
- Germany (3):
  - Charité Universitätsmedizin Berlin, Berlin
  - Asklepios Klinik Altona, Hamburg
  - Universitätsklinikum Ulm, Ulm
- Latvia (2):
  - Pauls Stradiņš Clinical University Hospital, Riga
  - Riga East Clinical University Hospital, Riga
- Lithuania (2):
  - The Hospital of Lithuanian University of Health Sciences, Kaunas
  - National Cancer Institute, Vilnius
- Netherlands (2):
  - Netherlands Cancer Institute, Amsterdam
  - Erasmus University Medical Center, Department of Medical Oncology, Rotterdam
- Oslo University Hospital, Radiumhospitalet, Oslo, Norway
- Spain (3):
  - Hospital 12 de Octubre, Madrid
  - Hospital Universitario Quirónsalud Madrid, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
- Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Paulus A, Zemaitis M, Cicenas S, Zvirbule Z, Sanfridson A, Millrud CR, Magnusson S, Losic N, Tersago D, Garcia-Ribas I, Thorsson L, Paz-Ares LG. Safety, efficacy, and analysis of biomarkers in patients with advanced non-small cell lung cancer treated with the anti-IL1RAP antibody nadunolimab (CAN04) in combination with platinum doublet. Lung Cancer. 2025 Aug;206:108664. doi: 10.1016/j.lungcan.2025.108664. Epub 2025 Jul 14. PMID 40680438
- [Derived] Robbrecht D, Jungels C, Sorensen MM, Spanggaard I, Eskens F, Fretland SO, Guren TK, Aftimos P, Liberg D, Svedman C, Thorsson L, Steeghs N, Awada A. First-in-human phase 1 dose-escalation study of CAN04, a first-in-class interleukin-1 receptor accessory protein (IL1RAP) antibody in patients with solid tumours. Br J Cancer. 2022 Apr;126(7):1010-1017. doi: 10.1038/s41416-021-01657-7. Epub 2021 Dec 13. PMID 34903842
- See also: Poster presentation at ESMO 2018 — https://cantargia.com/assets/uploads/Poster-CANFOUR-ESMO-2018-version-FINAL.pdf
- See also: Oral presentation at ASCO annual meeting 2019 — https://cantargia.com/assets/uploads/ASCO2019_CANFOUR-Phase-I_FINAL-01June_2019.pdf
- See also: Poster presentation at ESMO 2021 — https://cantargia.com/assets/uploads/538P-Awada-et-al-ESMO-2021.pdf
- See also: Poster presentation at ASCO annual meeting 2022 — https://cantargia.com/assets/uploads/Cantargia-ASCO-2022-Poster-9020-CANFOUR-NSCLC.pdf
- See also: Poster presentation at ASCO annual meeting 2022 — https://cantargia.com/assets/uploads/Cantargia-ASCO-2022-Poster-4141-CANFOUR-PDAC.pdf
- See also: Poster presentation at AACR annual meeting 2023 — https://cantargia.com/assets/uploads/AACR-2023-PDAC-poster.pdf
- See also: Poster presentation at ASCO annual meeting 2023 — https://cantargia.com/assets/uploads/ASCO-2023-NSCLC-poster.pdf